CLINICAL TRIAL: NCT03039114
Title: An Open-Label, Dose-Finding, and Cohort-Expansion Phase 1 Study Evaluating Safety and Efficacy of INCB050465 in Combination With Bendamustine and Obinutuzumab in Subjects With Relapsed or Refractory Follicular Lymphoma (CITADEL-102)
Brief Title: Study Evaluating Safety and Efficacy of INCB050465 Combined With Bendamustine and Obinutuzumab in Relapsed or Refractory Follicular Lymphoma (CITADEL-102)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 50465-102 (CITADEL-102); Parsaclisib (Other: Incyte Corporation); 2016-002829-11 (EudraCT Number)
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma
Keywords: Follicular lymphoma; relapsed; refractory; non-Hodgkin lymphoma; phosphatidylinositol 3-kinase (PI3K)
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Recurrence; Lymphoma, Non-Hodgkin | interventions — parsaclisib; Bendamustine Hydrochloride; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Parsaclisib + Hexal and Gazyvaro (Experimental)
  Interventions: Drug: Parsaclisib; Drug: Hexal; Drug: Gazyvaro

INTERVENTIONS:
Drug: Parsaclisib — Parsaclisib at the protocol-defined starting dose administered once daily for 8 weeks followed by once weekly.
  Other Names: INCB050465
Drug: Hexal — Bendamustine 90 mg/m^2 administered intravenously at protocol-defined timepoints.
  Other Names: Bendamustine
Drug: Gazyvaro — Obinutuzumab 1000 mg by intravenous infusion at protocol-defined timepoints.
  Other Names: Gazyva®; Obinutuzumab

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of parsaclisib when combined with bendamustine and obinutuzumab in subjects with relapsed or refractory follicular lymphoma (FL).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed FL.
* Documented CD20+ FL.
* Relapsed or refractory to any prior rituximab-containing regimen.
* Previously treated with a maximum of 4 cancer-directed treatment regimens.
* At least 1 measurable lesion > 1.5 cm in at least 1 dimension by computed tomography or magnetic resonance imaging.
* Must be willing to undergo an incisional or excisional lymph node biopsy of accessible adenopathy or provide the most recent, available archived tumor biopsy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.

Exclusion Criteria:

* Clinical evidence of transformation to a more aggressive subtype of lymphoma or Grade 3B FL.
* History of central nervous system lymphoma (either primary or metastatic).
* Allogeneic stem cell transplant within the last 6 months, or active graft-versus-host disease following allogeneic transplant or autologous stem cell transplant within the last 3 months before the date of the first dose of study drug administration.
* Use of any potent cytochrome P450 3A4 inhibitors or inducers within 14 days or 5 half-lives (whichever is longer) before the first dose of study drug.
* Prior treatment with a selective PI3Kδ inhibitor or a pan PI3K inhibitor.
* Prior treatment with bendamustine (within 12 months of the start of study treatment). Subjects with prior bendamustine treatment (> 12 months before the start of study treatment) are eligible if they meet the following criteria:

  * Did not discontinue because of tolerability concerns.
  * Achieved either partial or CR to the bendamustine regimen of at least 12 months in duration before relapse/progression.
  * Experienced progression following a regimen containing an alkylating agent.
* Received prior obinutuzumab.
* Received rituximab within 4 weeks of study start.
* Prior treatment-related toxicities that have not resolved to ≤ Grade 1 before the date of study drug administration except for stable chronic toxicities (≤ Grade 2) not expected to resolve (eg, stable Grade 2 peripheral neurotoxicity).
* Received any prior monoclonal antibody (except an anti-CD20 antibody) within 90 days before the date of study start.
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (eg, subjects in whom re-administration with rituximab would be contraindicated for safety reasons).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of parsaclisib in combination with bendamustine and obinutuzumab in relapsed or refractory FL, assessed by number of subjects with adverse events (AEs) | Screening through 30-35 days after end of treatment, up to approximately 34 months per subject

SECONDARY OUTCOMES:
Objective response rate based on Lugano classification criteria | Protocol-defined timepoints throughout the treatment period, up to approximately 34 months per subject
  Defined as percentage of subjects with a complete response (CR) and partial response (PR), as determined by investigator assessment of response
Complete response rate based on Lugano classification criteria | Protocol-defined timepoints throughout the treatment period, up to approximately 34 months per subject
  Defined as percentage of subjects who achieve a best overall response of CR
Duration of response | Protocol-defined timepoints throughout the treatment period, up to approximately 34 months per subject
  Defined as time from first documented evidence of CR or PR until earliest date of disease progression or death due to any cause.
Progression-free survival | Protocol-defined timepoints throughout the treatment period, up to approximately 34 months per subject
  Defined as time from the date of the first dose of study drug until the earliest date of disease progression (determined by radiographic disease assessment/Lugano classification criteria) or death due to any cause.
Overall survival | From the date of the first dose of study drug until death due to any cause, assessed up to approximately 34 months per subject
  Defined as the time from the date of the first dose of study drug until death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Fitzroy Dawkins, MD, Study Director — Incyte Corporation
Locations (21):
- United States (6):
  - Banner Health, Gilbert, Arizona
  - University of California, San Diego, La Jolla, California
  - University of Kansas Cancer Center, Fairway, Kansas
  - Center for Cancer and Blood Disorders (CCBD) - Bethesda, Bethesda, Maryland
  - Clinical Research Alliance, Lake Success, New York
  - Froedtert & Medical College of Wisconsin & Affiliated Hospitals, Milwaukee, Wisconsin
- FN Ostrava / Ostrava, Ostrava, Czechia
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - The Finsen Centre, National Hospital, Copenhagen
- Semmelweis Egyetem, Budapest, Hungary
- Italy (5):
  - Centro di Riferimento Oncologico, Aviano
  - Azienda Ospedaliero Universitaria Di Bologna, Bologna
  - Policlinico S. Orsola-Ematologia LA Seragnoli, Bologna
  - A.O. Spedali Civili, Brescia
  - UO Ematologia ASST Spedali Civili, Brescia
- Spain (5):
  - Hospital Germans Trias Pujol, Barcelona
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: Undecided